CLINICAL TRIAL: NCT02466971
Title: A Randomized Phase III Trial of Radiation Therapy and Cisplatin Alone or in Combination With Intravenous Triapine in Women With Newly Diagnosed Bulky Stage IB2, Stage II, IIIB, or IVA Cancer of the Uterine Cervix or Stage II-IVA Vaginal Cancer
Brief Title: Testing the Addition of a New Anti-Cancer Drug, Triapine, to the Usual Chemotherapy Treatment (Cisplatin) During Radiation Therapy for Advanced-stage Cervical and Vaginal Cancers
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00835; NCI-2015-00835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY006; NRG-GY006 (Other: NRG Oncology); NRG-GY006 (Other: CTEP); U10CA180868 (NIH); NCT01835171 (obsolete NCT alias); NCT05358600 (obsolete NCT alias)
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Results first posted 2024-01-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-07

CONDITIONS: Advanced Vaginal Adenocarcinoma; Advanced Vaginal Adenosquamous Carcinoma; Advanced Vaginal Squamous Cell Carcinoma; Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Squamous Cell Carcinoma; Stage IB2 Cervical Cancer AJCC v6 and v7; Stage II Cervical Cancer AJCC v7; Stage II Vaginal Cancer AJCC v6 and v7; Stage IIA Cervical Cancer AJCC v7; Stage IIB Cervical Cancer AJCC v6 and v7; Stage III Vaginal Cancer AJCC v6 and v7; Stage IIIB Cervical Cancer AJCC v6 and v7; Stage IV Vaginal Cancer AJCC v6 and v7; Stage IVA Cervical Cancer AJCC v6 and v7; Stage IVA Vaginal Cancer AJCC v6 and v7; Unresectable Vaginal Carcinoma; Vaginal Adenocarcinoma; Vaginal Adenosquamous Carcinoma; Vaginal Carcinoma; Vaginal Squamous Cell Carcinoma, Not Otherwise Specified
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms | interventions — Brachytherapy; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Congresses as Topic; Radiation; Radiotherapy, Intensity-Modulated; Radiotherapy; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (cisplatin, IMRT or RT, brachytherapy) (Active Comparator): Patients receive cisplatin IV over 90 minutes on days 2, 9, 16, 23, 30, (and day 36 or 37 at the treating physician's discretion). Patients then undergo EBRT (either conventional RT or IMRT) QD 5 days a week for 25 fractions followed by LDR or HDR brachytherapy according to institution's standards. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Brachytherapy; Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy
- Arm II (cisplatin, IMRT or RT, brachytherapy, triapine) (Experimental): Patients receive cisplatin and undergo EBRT followed by brachytherapy as in Arm I. Patients also receive triapine IV over 2 hours on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Brachytherapy; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy; Drug: Triapine

INTERVENTIONS:
Radiation: Brachytherapy — Undergo brachytherapy
  Other Names: Brachytherapy, NOS; Internal Radiation; Internal Radiation Brachytherapy; Internal Radiation Therapy; Radiation Brachytherapy; Radiation, Internal
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
  Arms: Arm I (cisplatin, IMRT or RT, brachytherapy)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radiation Therapy — Undergo conventional RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Triapine — Given IV
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811
  Arms: Arm II (cisplatin, IMRT or RT, brachytherapy, triapine)

SUMMARY:
This randomized phase III trial studies radiation therapy and cisplatin with triapine to see how well they work compared to the standard radiation therapy and cisplatin alone in treating patients with newly diagnosed stage IB2, II, or IIIB-IVA cervical cancer or stage II-IVA vaginal cancer. Radiation therapy uses high energy protons to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Triapine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether radiation therapy and cisplatin are more effective with triapine in treating cervical or vaginal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the efficacy of the experimental regimen of triapine (3AP), cisplatin, and radiation to increase overall survival relative to the standard/control regimen of cisplatin and radiation in women with uterine cervix or vaginal cancer.

SECONDARY OBJECTIVE:

I. To determine the relative progression-free survival impact of triapine-cisplatin radio-chemotherapy and cisplatin radio-chemotherapy.

TERTIARY OBJECTIVES:

I. To evaluate incidence and severity of hematologic and gastrointestinal (GI) adverse events by radiation modality; image guided intensity modulated radiation therapy (IG-IMRT) versus conventional pelvic radiotherapy. (05/30/2017) II. To summarize and compare differences in acute adverse events (Common Terminology Criteria for Adverse Events [CTCAE], version [v]4.0) by treatment arm and by radiation modality. (05/30/2017) III. To summarize and compare differences in chronic or late (>= 30-days from off study treatment date) adverse events (CTCAE, v4.0) by treatment arm and by radiation modality. (05/30/2017) IV. To determine peripheral blood methemoglobin proportion before and after triapine infusion (optional for Arm 2 patients).

V. To explore whether knowledge-based planning (KBP) can improve IG-IMRT plans compared to plans that would have been delivered without KBP, estimate the resulting toxicity reduction using normal tissue complication probability (NTCP) models, and determine whether KBP should be a requirement for future IG-IMRT protocols.

VI. To determine the post-therapy 3-month fludeoxyglucose F-18 (18F-FDG) PET/CT metabolic complete response rate by treatment arm VII. To compare acute toxicity and chemotherapy delivery for atlas-based IG-IMRT vs. positron emission tomography (PET)/computed tomography (CT)-based IG-IMRT vs. conventional radiation therapy (RT), and assess the impact of treatment on changes in hematopoietic compensatory response.

VIII. To develop and validate machine learning and radiomics techniques for dose accumulation, automated treatment planning, and prediction of treatment response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive cisplatin intravenously (IV) over 90 minutes on days 2, 9, 16, 23, 30, (and day 36 or 37 at the treating physician's discretion). Patients then undergo external beam radiation therapy (EBRT) (either conventional RT or intensity modulated radiation therapy [IMRT]) once daily (QD) 5 days a week for 25 fractions followed by low dose rate (LDR) or high dose rate (HDR) brachytherapy according to institution's standards. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cisplatin and undergo EBRT followed by brachytherapy as in Arm I. Patients also receive triapine IV over 2 hours on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 and 3 months, every 3 months for 2 years, and then every 6 months for 3 years.

The patient data from NCI #9434 will be merged with NRG-GY006 per the Protocol Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a new, unrated histologic diagnosis of stage IB2 (> 4 cm), II, IIIB or IVA squamous, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix (FIGO 2009) or stage II-IVA squamous, adenocarcinoma, or adenosquamous carcinoma of the vagina not amenable to curative surgical resection alone; the presence or absence of para-aortic lymph node metastasis will be based on pre-therapy 18F-FDG PET/CT; NOTE: if the baseline 18F-FDG PET/CT identifies hypermetabolic para-aortic disease, such patients will NOT be eligible; the patient must be able to tolerate imaging requirements of an 18F-FDG PET/CT scan
* Patient must provide study specific informed consent prior to study entry
* Patient must have a Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2 or equivalent
* Absolute neutrophil count > 1,500/uL
* Platelets > 100,000/uL
* Hemoglobin > 10 g/dL
* Total bilirubin < 2.0 mg/dL
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal
* Prothrombin time (PT)/activated partial thromboplastin time (aPTT) < 1.5 X institutional upper limit of normal
* Creatinine =< 1.5 mg/dL to receive weekly cisplatin

  * Patients whose serum creatinine is between 1.5 and 1.9 mg/dL are eligible for cisplatin if the estimated creatinine clearance (CCr) is >= 30 ml/min; for the purpose of estimating the CCr, the formula of Cockcroft and Gault for females should be used
* Patient does not have uncontrolled diabetes mellitus (i.e., fasting blood glucose > 200 mg/dL)
* Patient has a life expectancy of greater than 20 weeks
* Patient does not have known brain metastases (testing optional)
* Patient does not have known human immunodeficiency virus syndrome (HIV, testing optional); known HIV-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with triapine
* Patient does not have a known allergy to compounds of similar or biologic composition as triapine
* Patient does not have known glucose-6-phosphate dehydrogenase (G6PD) deficiency as the condition interferes with triapine antidote metabolism (G6PD testing optional)
* Patient is not actively breastfeeding (or has agreed to discontinue breastfeeding before the initiation of protocol therapy)

Exclusion Criteria:

* Patient has another concurrent active invasive malignancy
* Patient has had a prior invasive malignancy diagnosed within the last three years (except [1] non-melanoma skin cancer or [2] prior in situ carcinoma of the cervix); patients are excluded if they have received prior pelvic radiotherapy for any reason that would contribute radiation dose that would exceed tolerance of normal tissues at the discretion of the treating physician
* Patient has uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within six months of protocol initiation, cardiac arrhythmia within six months of protocol initiation; known inadequately controlled hypertension; clinically significant pulmonary disease including dyspnea at rest, or patients requiring supplemental oxygen, or poor pulmonary reserve; or clinically significant renal function impairment (baseline serum creatinine > 2 mg/dL); or psychiatric illness/social situations that would limit compliance with study requirements
* Patient is receiving another investigational agent for the treatment of cancer
* Patient is currently pregnant
* Patient does not agree to use two forms of birth control if they are of child-bearing potential
* Patients who have had a hysterectomy or are planning to have an adjuvant hysterectomy following radiation as part of their cervical cancer treatment are ineligible (05/30/2017)
* Patients scheduled to be treated with adjuvant consolidation chemotherapy or other anti-neoplastic therapy at the conclusion of their standard chemoradiation (05/30/2017)
* Patients with self-reported or known diagnosis of G6PD deficiency (05/30/2017)
* Patients with vaginal cancer may have previously undergone a hysterectomy for various indications; patients with vaginal cancer who underwent a hysterectomy for treatment of cervical cancer less than five years prior to their diagnosis of vaginal cancer are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2026-07-14 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Leath, Principal Investigator — NRG Oncology
Locations (382):
- United States (378):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Cooper CyberKnife Center, Mount Laurel, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Saint Peter's Health Partners, Albany, New York
  - Women's Cancer Care Associates LLC, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- Puerto Rico (3):
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Kunos CA, Andrews SJ, Moore KN, Chon HS, Ivy SP. Randomized Phase II Trial of Triapine-Cisplatin-Radiotherapy for Locally Advanced Stage Uterine Cervix or Vaginal Cancers. Front Oncol. 2019 Oct 15;9:1067. doi: 10.3389/fonc.2019.01067. eCollection 2019. PMID 31681600
- [Derived] Kunos CA, Ivy SP. Triapine Radiochemotherapy in Advanced Stage Cervical Cancer. Front Oncol. 2018 May 7;8:149. doi: 10.3389/fonc.2018.00149. eCollection 2018. PMID 29868473

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NRG-GY006 opened to accrual on January 15, 2016, and closed to accrual on September 22, 2022.
Period: Overall Study
Arm/Group | Arm I (Cisplatin, IMRT or RT, Brachytherapy) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine)
Started | 225 | 225
Completed | 207 | 202
Not Completed | 18 | 23
Not completed — eligible and never treated | 14 | 20
Not completed — too early for evaluation of treatment and toxicity | 3 | 2
Not completed — ineligible and treated | 1 | 0
Not completed — ineligible and never treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cisplatin, IMRT or RT, Brachytherapy) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine) | Total
Number analyzed (Participants) | 224 | 224 | 448
Age, Continuous [Median (Full Range); unit: years] | 47 [23 to 82] | 47 [26 to 85] | 47 [23 to 85]
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 7 | 8 | 15
  30-39 years | 58 | 50 | 108
  40-49 years | 64 | 73 | 137
  50-59 years | 57 | 49 | 106
  60-69 years | 27 | 27 | 54
  70-79 years | 9 | 13 | 22
  >= 80 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 224 | 448
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 57 | 101
  Not Hispanic or Latino | 169 | 164 | 333
  Unknown or Not Reported | 11 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 10
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 32 | 36 | 68
  White | 165 | 160 | 325
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate at 3 Years
Description: Estimate for probability of overall survival at 3 years by Kaplan-Meier method, where overall survival is defined as the time from randomization to time of death due to any cause or the date of last contact, whichever occurs first.
Time Frame: At 3 years from randomization.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Cisplatin, IMRT or RT, Brachytherapy) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine)
Number analyzed (Participants) | 224 | 224
percentage of participants | 78.1 [70 to 84] | 79.6 [72 to 85]

2. Secondary Outcome: Progression-free Survival (PFS) Rate at 3 Years
Description: Estimate for probability of progression free at 3 years by Kaplan-Meier method, where progression-free survival is defined as the time from randomization to the date of first documented disease recurrence/progression, death from any cause or date of last contact, whichever occurs first. Recurrence is defined as clinical, radiological or histological evidence of recurrent disease post study treatment. Disease progression will be determined from the physical examinations, which were conducted during treatment (day 9, 16, 23, 30 and 37) and follow-up (1 and 3 months after completing protocol therapy, every 3 months for years 1 and 2, and every 6 months for years 3, 4 and 5), and the PET/CT scan conducted 3 months after the end of treatment. Please note that progression defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1) is not required by the protocol.
Time Frame: At 3 years from study randomization.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Cisplatin, IMRT or RT, Brachytherapy) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine)
Number analyzed (Participants) | 224 | 224
percentage of participants | 69.5 [62 to 76] | 71.4 [64 to 78]

3. Secondary Outcome: Number of Participants With Adverse Events (Grade 3 or Higher) During Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: During treatment period and up to 30 days after stopping the study treatment with a median treatment time as 53 days ranging from 1 to 189 days.
Population: Participants who received any study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Cisplatin, IMRT or RT, Brachytherapy) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine)
Number analyzed (Participants) | 208 | 202
Participants
  Anemia | 23 | 18
  Other blood and lymphatic system disorders | 5 | 7
  White blood cell count decreased | 19 | 17
  Platelet count decreased | 5 | 2
  Neutrophil count decreased | 13 | 4
  Other investigations | 39 | 41
  Cardiac disorders | 0 | 2
  Eye disorders | 0 | 1
  Gastrointestinal disorders | 22 | 22
  General disorders | 7 | 1
  Hepatobiliary disorders | 1 | 0
  Infections and infestations | 17 | 12
  Metabolism and nutrition disorders | 29 | 22
  Musculoskeletal and connective tissue disorders | 2 | 3
  Neoplasms benign, malignant and unspecified | 0 | 1
  Nervous system disorders | 5 | 4
  Psychiatric disorders | 1 | 1
  Renal and urinary disorders | 3 | 4
  Reproductive system and breast disorders | 8 | 11
  Respiratory, thoracic and mediastinal disorders | 0 | 1
  Skin and subcutaneous tissue disorders | 1 | 0
  Surgical and medical procedures | 1 | 0
  Vascular disorders | 20 | 11

4. Other Pre Specified Outcome: Number of Participants With Hematologic Toxicity During Treatment Period
Description: Number of participants with hematologic toxicity during treatment period, where hematologic toxicity is defined as occurrence of any grade 3 or higher adverse events for neutropenia, leukopenia, lymphopenia, anemia, or thrombocytopenia. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: Up to 30 days after completion of study treatment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Participants With Adverse Events (Grade 3 or Higher) That Occurred During Follow-Up Period
Description: Number of participants with a maximum grade of 3 or higher that occurred during follow-up period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Peripheral Blood Methemoglobin
Description: Peripheral blood methemoglobin collected at baseline and 1, 3, 5 and 24 hours after Triapine infusion on Day 1 in Arm II.
Time Frame: Baseline to 24 hours after triapine infusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Metabolic Complete Response (mCR)
Description: The assessment of metabolic complete response is based on the ratio of post 3-month therapy PET/CT maximum standardized update value (SUV) to pre-therapy PET/CT maximum SUV. The metabolic complete response is classified as complete response for a ratio of 0.33 or less, or partial response for a ratio between 0.34 and 0.75, or stable response for a ratio greater that 0.75 but less than 1.25, or progressive response for a ratio greater than 1.25.
Time Frame: Up to 3 months after completion of treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Intensity Modulated Radiation Therapy (IG-IMRT)
Description: Number of Participants with KBP IG-IMRT
Time Frame: Up to 60 days.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment period (median: 53 days) and up to 30 days after stopping the study treatment for participants who received any study treatment. All-cause mortality that occurred through study completion with a median follow-up as 28 months (inter-quartile range: 15 to 45 months) by reverse Kaplan-Meier method.
Description: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment for participants who received any study treatment. Note that the population is different for all-cause mortality and adverse events. For all-cause mortality the population is "all eligible participants." For adverse event reporting, the population is "all patients who received any study treatment."
Arm/Group | Arm I (Cisplatin, IMRT or RT, Brachytherapy) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine)
All-Cause Mortality (participants affected / at risk) | 35/224 | 34/224
Serious Adverse Events (participants affected / at risk) | 45/208 | 45/202
Other Adverse Events (participants affected / at risk) | 198/208 | 194/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cisplatin, IMRT or RT, Brachytherapy) (N=208) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine) (N=202)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 6 | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Chest Pain - Cardiac (Cardiac disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 2
Duodenal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 0
General Disorders And Administration Site Conditio (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 4 | 0
Infections And Infestations - Other (Infections and infestations) | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Kidney Infection (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 4 | 1
Appendicitis (Infections and infestations) | 0 | 1
Uterine Perforation (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 1
White Blood Cell Decreased (Investigations) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
Thromboembolic Event (Vascular disorders) | 4 | 4
Hypertension (Vascular disorders) | 4 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Cisplatin, IMRT or RT, Brachytherapy) (N=208) | Arm II (Cisplatin, IMRT or RT, Brachytherapy, Triapine) (N=202)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 | 1
Lymph Node Pain (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 2 | 4
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1 | 2
Anemia (Blood and lymphatic system disorders) | 105 | 105
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Atrial Fibrillation (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 7
Cardiac Disorders - Other (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 8 | 12
Chest Pain - Cardiac (Cardiac disorders) | 0 | 2
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 2 | 3
Vertigo (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 45 | 21
Hearing Impaired (Ear and labyrinth disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0
Endocrine Disorders - Other (Endocrine disorders) | 1 | 2
Eye Disorders - Other (Eye disorders) | 0 | 2
Watering Eyes (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 0 | 2
Glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1
Blurred Vision (Eye disorders) | 6 | 6
Dry Eye (Eye disorders) | 1 | 1
Floaters (Eye disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 14 | 22
Dry Mouth (Gastrointestinal disorders) | 3 | 4
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 64 | 73
Diarrhea (Gastrointestinal disorders) | 144 | 139
Vomiting (Gastrointestinal disorders) | 60 | 55
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 6 | 5
Duodenal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Stomach Pain (Gastrointestinal disorders) | 5 | 9
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Anal Mucositis (Gastrointestinal disorders) | 0 | 1
Rectal Fistula (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 44 | 50
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 6 | 7
Mucositis Oral (Gastrointestinal disorders) | 9 | 9
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 9 | 5
Anal Pain (Gastrointestinal disorders) | 2 | 3
Oral Hemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 141 | 126
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 16 | 15
Rectal Pain (Gastrointestinal disorders) | 8 | 4
Fecal Incontinence (Gastrointestinal disorders) | 0 | 2
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 2 | 5
Toothache (Gastrointestinal disorders) | 2 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 5 | 5
Gastritis (Gastrointestinal disorders) | 2 | 2
General Disorders And Administration Site Conditio (General disorders) | 7 | 13
Pain (General disorders) | 14 | 25
Malaise (General disorders) | 2 | 2
Localized Edema (General disorders) | 5 | 0
Flu Like Symptoms (General disorders) | 2 | 2
Edema Trunk (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 5 | 15
Edema Limbs (General disorders) | 10 | 17
Facial Pain (General disorders) | 0 | 1
Edema Face (General disorders) | 1 | 3
Fatigue (General disorders) | 122 | 120
Fever (General disorders) | 15 | 19
Chills (General disorders) | 9 | 7
Infusion Related Reaction (General disorders) | 1 | 3
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Allergic Reaction (Immune system disorders) | 2 | 1
Infections And Infestations - Other (Infections and infestations) | 6 | 13
Wound Infection (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 1
Tooth Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 2 | 6
Sinusitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 3
Rash Pustular (Infections and infestations) | 0 | 1
Peripheral Nerve Infection (Infections and infestations) | 1 | 0
Papulopustular Rash (Infections and infestations) | 1 | 2
Mucosal Infection (Infections and infestations) | 0 | 2
Lung Infection (Infections and infestations) | 1 | 2
Kidney Infection (Infections and infestations) | 4 | 1
Device Related Infection (Infections and infestations) | 1 | 1
Vaginal Infection (Infections and infestations) | 1 | 3
Urinary Tract Infection (Infections and infestations) | 41 | 36
Lip Infection (Infections and infestations) | 1 | 0
Abdominal Infection (Infections and infestations) | 1 | 0
Injury, Poisoning And Procedural Complications - O (Injury, poisoning and procedural complications) | 0 | 1
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 | 1
Uterine Perforation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Dermatitis Radiation (Injury, poisoning and procedural complications) | 6 | 19
Burn (Injury, poisoning and procedural complications) | 0 | 2
Bruising (Injury, poisoning and procedural complications) | 8 | 5
Investigations - Other (Investigations) | 5 | 5
Weight Loss (Investigations) | 18 | 8
Weight Gain (Investigations) | 2 | 2
Platelet Count Decreased (Investigations) | 69 | 74
Lymphocyte Count Decreased (Investigations) | 48 | 51
Inr Increased (Investigations) | 1 | 1
Ggt Increased (Investigations) | 4 | 2
Creatinine Increased (Investigations) | 35 | 17
Cholesterol High (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 37 | 28
Cd4 Lymphocytes Decreased (Investigations) | 1 | 0
Blood Bilirubin Increased (Investigations) | 4 | 4
White Blood Cell Decreased (Investigations) | 88 | 75
Aspartate Aminotransferase Increased (Investigations) | 15 | 15
Alkaline Phosphatase Increased (Investigations) | 14 | 14
Alanine Aminotransferase Increased (Investigations) | 29 | 22
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 7 | 2
Obesity (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 7
Hyponatremia (Metabolism and nutrition disorders) | 48 | 41
Hypomagnesemia (Metabolism and nutrition disorders) | 69 | 60
Hypokalemia (Metabolism and nutrition disorders) | 47 | 38
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 37 | 38
Hypoalbuminemia (Metabolism and nutrition disorders) | 46 | 45
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 10 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 45 | 44
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 9
Glucose Intolerance (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 16 | 14
Anorexia (Metabolism and nutrition disorders) | 47 | 45
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 | 12
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle Weakness Left-Sided (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 8 | 5
Flank Pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 24 | 23
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Musculoskeletal And Connective Tissue Disorder - O (Musculoskeletal and connective tissue disorders) | 10 | 8
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nervous System Disorders - Other (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 3 | 5
Stroke (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 20 | 10
Peripheral Motor Neuropathy (Nervous system disorders) | 2 | 0
Paresthesia (Nervous system disorders) | 5 | 2
Neuralgia (Nervous system disorders) | 0 | 3
Memory Impairment (Nervous system disorders) | 1 | 3
Lethargy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 53 | 46
Encephalopathy (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 21 | 19
Sinus Pain (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 2
Dizziness (Nervous system disorders) | 33 | 29
Concentration Impairment (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Psychiatric Disorders - Other (Psychiatric disorders) | 1 | 2
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Libido Decreased (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 23 | 33
Depression (Psychiatric disorders) | 10 | 11
Delirium (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 23 | 28
Agitation (Psychiatric disorders) | 5 | 3
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 20 | 19
Urinary Urgency (Renal and urinary disorders) | 12 | 15
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 3 | 2
Urinary Incontinence (Renal and urinary disorders) | 5 | 9
Urinary Tract Pain (Renal and urinary disorders) | 16 | 23
Urinary Frequency (Renal and urinary disorders) | 32 | 40
Urinary Fistula (Renal and urinary disorders) | 0 | 1
Renal Calculi (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 14 | 11
Hematuria (Renal and urinary disorders) | 14 | 15
Cystitis Noninfective (Renal and urinary disorders) | 23 | 36
Bladder Spasm (Renal and urinary disorders) | 0 | 2
Acute Kidney Injury (Renal and urinary disorders) | 3 | 3
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 4 | 6
Vaginal Perforation (Reproductive system and breast disorders) | 0 | 1
Vaginal Pain (Reproductive system and breast disorders) | 8 | 9
Vaginal Hemorrhage (Reproductive system and breast disorders) | 52 | 45
Vaginal Fistula (Reproductive system and breast disorders) | 1 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1
Uterine Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Premature Menopause (Reproductive system and breast disorders) | 0 | 1
Perineal Pain (Reproductive system and breast disorders) | 1 | 1
Pelvic Pain (Reproductive system and breast disorders) | 39 | 29
Menorrhagia (Reproductive system and breast disorders) | 3 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 25 | 32
Vaginal Inflammation (Reproductive system and breast disorders) | 2 | 5
Genital Edema (Reproductive system and breast disorders) | 0 | 1
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 2 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 0
Breast Pain (Reproductive system and breast disorders) | 0 | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 15 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 5 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5
Periorbital Edema (Skin and subcutaneous tissue disorders) | 0 | 1
Pain Of Skin (Skin and subcutaneous tissue disorders) | 2 | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 9 | 8
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Ridging (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 5 | 8
Body Odor (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 8
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 2 | 1
Vascular Disorders - Other (Vascular disorders) | 1 | 1
Thromboembolic Event (Vascular disorders) | 8 | 9
Superficial Thrombophlebitis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 7
Hypertension (Vascular disorders) | 25 | 22
Hot Flashes (Vascular disorders) | 28 | 19
Hematoma (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT02466971/Prot_SAP_001.pdf